CLINICAL TRIAL: NCT00786058
Title: A Phase III Second Line Trial of Patients With Gemcitabine Resistant Advanced Pancreatic Cancer (CONKO-003)
Brief Title: A Phase III Second Line Trial in Advanced Pancreatic Cancer CONKO 003
Status: Approved for marketing | Type: Expanded Access
Sponsor: CONKO-Studiengruppe (Other)
Collaborators: Sanofi (Industry); medac GmbH (Industry); Amgen (Industry)
Responsible Party: Helmut Oettle PHD, CONKO Study group
Other Study IDs: CONKO 003; CCT-NAPN-16751
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Pancreatic Cancer
Keywords: refractory pancreatic cancer; gemcitabine; phase III; second line
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Fluorouracil

INTERVENTIONS:
Drug: OFF in experimental arm — OFF was given according to a six week cycle. FA (500 mg/m2 , 0.5h, i.v.) and 5-FU (2,600 mg/m2, 24-hour, i.v.) were administered on days 1, 8, 15, and 22. Oxaliplatin (85 mg/m2 , 2-4 h, i.v.) was administered directly before FA/ 5-FU on days 8 and 22.
  Other Names: Eloxatin; Calciumfolinat; 5-Fluorouracil

SUMMARY:
The purpose of this study is to compare best supportive care plus oxaliplatin/ folinic acid/ 5-FU versus best supportive alone in patients with gemcitabine refractory pancreatic cancer.

DETAILED DESCRIPTION:
Gemcitabine (G) given until progressive disease (PD) is still standard therapy in patients with advanced pancreatic cancer. No standard secondline regimen is available after PD. Best supportive care (BSC) is the main option for these patients. Our phase II study (Pelzer et al, ASCO 2002) showed activity of the OFF (Oxaliplatin/Folinic Acid/5-FU) regimen. To confirm these data we started this multicenter phase III study to examine OFF vs. BSC alone.

165 patients were needed for this study. Following CT/ MRT confirmed PD patients were randomized. Stratification included duration of firstline therapy, Karnofsky Performance Status (KPS) and tumor stage. OFF (outpatient regimen): 5-FU 2g/m² (24h)/FA 200 mg/m² (30min) on d1, d8, d15, d22, additional Oxaliplatin 85mg/m² (2h) on day 8 and 22. Rest on day 23 and 42.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic pancreatic adenocarcinoma that had progressed during first line gemcitabine therapy were eligible for inclusion in the study.

Other inclusion criteria were:

* Age > 18 years
* Karnofsky performance status > 70%
* Bidimensionally measurable reference lesion, adequate laboratory values for hematology (white blood cell [WBC] count > 3.5´109/L, platelet count > 100´109/L), renal function (creatine clearance > 30 ml/min) and hepatic function (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] < 2.5 ´ upper normal limit [UNL] and in the case of liver metastasis < 5 x UNL)
* As well as controlled pain

Exclusion Criteria:

* Patients were excluded from the study if they had any severe concurrent medical condition interfering with planned therapy, serious cardiac disease, sensory/ motor neuropathy > grade 2 or had previous or current malignancies at other origin; besides, pregnant or lactating women were excluded.
* All patients provided written informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Oettle, PD, Principal Investigator — CONKO Study Group

REFERENCES:
- [Derived] Oettle H, Riess H, Stieler JM, Heil G, Schwaner I, Seraphin J, Gorner M, Molle M, Greten TF, Lakner V, Bischoff S, Sinn M, Dorken B, Pelzer U. Second-line oxaliplatin, folinic acid, and fluorouracil versus folinic acid and fluorouracil alone for gemcitabine-refractory pancreatic cancer: outcomes from the CONKO-003 trial. J Clin Oncol. 2014 Aug 10;32(23):2423-9. doi: 10.1200/JCO.2013.53.6995. Epub 2014 Jun 30. PMID 24982456
- See also: Related Info — http://www.accessdata.fda.gov/scripts/cder/drugsatfda